CLINICAL TRIAL: NCT01448395
Title: An Open Label Single-Dose Study in Healthy Male Subjects Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]NXL104
Brief Title: Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]NXL104
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D4280C00008
Record Dates: First submitted 2011-09-30; First posted 2011-10-07 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Mass Balance; Metabolite Identification and Profiling; Metabolite profile and Identification of [14C]NXL104; Mass Balance Recovery

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: [14C]NXL104

INTERVENTIONS:
Drug: [14C]NXL104 — 500mg/100mL intravenous solution

SUMMARY:
A study to look at how radiolabelled NXL104 is taken up, broken down and removed by the body when given as an injection into the blood stream.

DETAILED DESCRIPTION:
An Open Label Single-Dose Study in Healthy Male Subjects Designed to Assess the Mass Balance Recovery, Metabolite profile and Metabolite Identification of [14C]NXL104.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Healthy male subjects aged 30-65 years inclusive.
* Male subjects should be willing to use an adequate method of contraception (as defined in Section 5.1) from the day of dosing until 3 months after dosing with the investigational product.
* Have a body mass index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg.
* Clinically normal physical examination and laboratory findings as judged by the investigator, including negative test results for drug abuse, alcohol, CO breath test and negative test results for Hepatitis B surface antigen, antibodies to Hepatitis C.

Exclusion Criteria:

* Any clinically significant disease or disorder (e.g. cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment).
* Any clinically relevant abnormal findings in physical examination, vital signs, clinical chemistry, haematology, urinalysis, which, in the opinion of the investigator, may put the subject at risk because of his participation in the study.
* QTc > 450 ms or QT > 500 ms or other ECG abnormality making interpretation more difficult, as judged by the investigator, or a history of additional risk factors for Torsades de Points (eg heart failure, hypokalemia, family history of long QT syndrome).
* Radiation exposure from clinical studies, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last twelve months or 10 mSv in the last five years.
* Participation in another clinical study with an investigational product during the last 3 months.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Mass balance after a single intravenous (IV) dose of [14C]NXL104 as generated from recovery of total radioactivity excreted in urine | 168 hours
Routes of [14C]NXL104 metabolism and excretion measured through total radioactivity concentrations in urine | 168 hours
Whole blood and plasma partitioning of total radioactivity through measurement of total radioactivy levels in blood | 168 hours
Mass balance after a single intravenous (IV) dose of [14C]NXL104 as generated from recovery of total radioactivity excreted in faeces | 168 hours
Routes of [14C]NXL104 metabolism and excretion measured through total radioactivity concentrations in faeces | 168 hours

SECONDARY OUTCOMES:
IV pharmacokinetics (PK) of [14C]NXL104 through calculation of Cmax, Tmax, AUC0-infinity, T1/2, MRT, terminal elimination rate constant, amount of NXL104 (Ae), % excreted, will be calculated from NXL104 concentrations in urine and faeces | Predose, 0.25, 0.5, 1,1.25,1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144, 168 hours
  Explanations for abbreviations:
  Cmax = Maximum concentration Tmax = Time taken to reach maximum concentration AUC 0-Infinity = Area under the plasma concentration-time curve 0-Infinity T1/2 = Terminal half-life MRT = Mean Residence Time
Metabolites of [14C]NXL104 in plasma, whole blood, urine and faeces calculated from plasma,urine and faces concentration levels.Identification of major metabolites in plasma,urine and faeces where possible | Whole blood:Predose, 0.25, 0.5, 1,1.25,1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144, 168 hoursUrine and Faeces samples Predose-144 hours
Safety and tolerability of NXL104 as number of patients with adverse events and assessment of Electrocardiogram (ECG) and vital signs results | Electrocardiogram (ECG) recordings at Screening Pre-dose, 1 ,24 and 168 hoursContinuous ECG monitoring 0-1 hourVital signs measurements screening pre-dose, 0.5, 1, 2, 24 and 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newell, MD, Study Director — AstraZeneca
Locations (1):
- Study site, Ruddington, Nottingham, United Kingdom

REFERENCES:
- See also: Redacted CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1454&filename=D4280C00008_CSP-Redacted.pdf